CLINICAL TRIAL: NCT05175222
Title: Assessment of Efficacy of LightWalker (Nd:Yag, Er:Yag) Laser Therapy on Incidence, Severity and Duration of Oral Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation (HSCT). Prospective Randomized Open-label Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOMOD-HSCT1
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Oral Mucositis; Bone Marrow Transplant Complications
Keywords: oral mucositis; low-level laser therapy; biomodulation; hematopoietic stem cell transplantation
MeSH Terms: conditions — Stomatitis | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Patients receive low-level laser therapy with LightWalker laser from the first day of conditioning chemotherapy till +2 day post hematopoietic stem cell transplantation. Additionally, standard supportive care is introduced.
  Interventions: Radiation: Laser therapy
- Control (No Intervention): Patients are observed and receive standard supportive care.

INTERVENTIONS:
Radiation: Laser therapy — Patients receive laser therapy in 7 points in oral cavity every day from the first day of conditioning chemotherapy till the second day post HSCT. Each point is irradiated for 1 minute.
  Arms: Laser

SUMMARY:
Oral mucositis (OM) is a common and debilitating adverse effect of conditioning regimens in patients undergoing hematopoietic cell transplantation (HCT). It is treated symptomatically with pain relief medications. The use of low-level laser therapy (LLLT) to prevent tissue damage has been postulated for almost forty years, however, there are only a few reports concerning old generation lasers in mucositis prophylaxis in HCT recipients. Here we hypothesized, that a new generation LLLT (Nd: YAG Fotona LightWalker®) laser may be an effective prophylaxis in shortening and reducing the severity of this complication.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized open-label study. All patients qualified to hematopoietic stem cell transplantation will be informed about possibility of taking part in this study. Patients who meet the inclusion criteria will be enrolled and randomized into two groups.

Patients in the first group will receive standard supportive treatment. Patients in the second group, except for the supportive treatment (as in the first group), will additionally receive prophylactic laser therapy of oral mucosa during high-dose chemotherapy conditioning before HSCT. Patients will undergo laser treatment daily from the first day of conditioning regimen till the second day after stem cell transfusion. The procedure will be carried out by trained staff at the bedside.

Severity of oral mucositis and pain will be measured in both groups on days 0, 4, 7, 11, 14, 18 and 21 after HSCT.

Severity of oral mucositis will be assessed according to five-point WHO scale Pain intensity will be measured on the basis of ten-point NRS scale.

In addition, the need for opioid analgesics and total parenteral nutrition will be evaluated.

Photographic documentation will be made on days -7, 0, 7, 14, 21. All obtained results will be collected in a database and subjected to statistical analysis. Additional analysis will be carried out during the study to evaluate whether the differences in results between studied groups reach statistical significance with less than a predetermined number of patients.

ELIGIBILITY:
Inclusion Criteria:

* written, informed consent for participation in the study
* oral sanation
* myeloablative conditioning

Exclusion Criteria:

* lack of patient's consent
* pathological lesions in oral cavity on the first day of conditioning regimen
* renal failure
* active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Duration of oral mucositis | First day of conditioning chemotherapy till 21 st day post hematopoietic stem cell transplantation
  Duration of oral mucositis duration in days measured in both groups
Severity of oral mucositis | First day of conditioning chemotherapy till 21 st day post hematopoietic stem cell transplantation
  Evaluation of pain according to NRS scale

SECONDARY OUTCOMES:
Need for opioid analgesics calculated | First day of conditioning chemotherapy till 21 st day post hematopoietic stem cell transplantation
  Opioid analgesic need assessed in days
Length of most severe pain | First day of conditioning chemotherapy till 21 st day post hematopoietic stem cell transplantation
  Number of days of most severe pain according to NRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Anna Irga-Staniukiewicz, MD, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code